CLINICAL TRIAL: NCT01282840
Title: Bladder Wall Blood Perfusion Pattern and Sexual Dysfunction in Female Patients With Lower Urinary Tract Symptoms, and the Association of That Perfusion Pattern and Therapeutic Efficacy of Antimuscarincs for Female Overactive Bladder Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 099049-F
Record Dates: First submitted 2011-01-23; First posted 2011-01-25 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2018-11

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: LUTS
MeSH Terms: conditions — Lower Urinary Tract Symptoms

ARMS (1):
- Bladder wall blood perfusion pattern (Other)
  Interventions: Drug: Tolterodine SR

INTERVENTIONS:
Drug: Tolterodine SR — Tolterodine SR 4 mg qd

SUMMARY:
Overactive bladder syndrome (OAB) affects around 17 % of female population. However, the etiology of OAB is complicated and unclear in many aspects. Bladder wall thickness had been reported to be strongly associated with OAB, but its use as a screening tool remains controversial. Besides, few studies reported patterns of sexual dysfunction in female patients with lower urinary tract symptoms (LUTS). Therefore the aims of our study were to analyze the bladder wall blood perfusion pattern in female LUTS patients, the association of between the bladder wall blood perfusion pattern and the efficacy of anti-muscarinic treatment for female OAB, and the patterns of sexual dysfunction in the female LUTS patients.

ELIGIBILITY:
Inclusion Criteria:

* all cases are female patients with lower urinary tract symptoms

Exclusion Criteria:

* nil

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2010-07-20 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Blood flow pattern after antimuscarinics | 12 weeks

SECONDARY OUTCOMES:
Blood flow patterns between different LUTS subgroups | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Banqiao, Taiwan